CLINICAL TRIAL: NCT07006168
Title: Effects Of Intra-Operative Intra-Articular Cocktail Injection In Patella Open Reduction And Internal Fixation (ORIF): A Single Centre, Double Blinded, Randomised Control Trial
Brief Title: Effects Of Intra-Operative Intra-Articular Cocktail Injection In Patella Open Reduction And Internal Fixation
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Christian Xinshuo Fang, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW 24-611
Record Dates: First submitted 2025-05-15; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-04

CONDITIONS: Patella Fracture
Keywords: Intra-Articular analgesic injection; Pain relief; Open Reduction and Internal Fixation; Functional Recovery; Rehabilitation; Range of motion; Post-operative recovery
MeSH Terms: conditions — Patella Fracture | interventions — Ketorolac; Triamcinolone Acetonide; Ropivacaine; Saline Solution; Epinephrine

STUDY DESIGN:
Intervention Model Description: Patients will be allocated to receive either Intra-articular Cocktail Injection (IA Cocktail) OR receive no Injection (Control).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intra-Articular Cocktail Injection (Experimental): After fixation, an intra-articular cocktail injection is injected into the surgical site. The intra-articular cocktail regime: Ketoralac 15mg, Ropivacaine 1% 15ml, 0.9% Normal Saline 35ml, Adrenaline 1:1000 0.5ml, Stacort-A Triamcinolone Acetonide 40mg. The total cocktail volume is approximately 50ml.
  Interventions: Drug: Ketorolac 15mg; Drug: Triamcinolone Acetonide 40mg; Drug: Ropivacaine HCL 1% 15ml; Drug: 0.9 % Normal Saline 35ml; Drug: Adrenaline 1:1000 0.5ml
- No Injection (No Intervention): No injection will be given to the patient.

INTERVENTIONS:
Drug: Ketorolac 15mg — An intra-articular cocktail injection ( Ketoralac 15mg, Ropivacaine 1% 15ml, 0.9% Normal Saline 35ml, Adrenaline 1:1000 0.5ml, Stacort-A Triamcinolone Acetonide 40mg) will be injected into the surgical site after fracture fixation surgery.
  Arms: Intra-Articular Cocktail Injection
Drug: Triamcinolone Acetonide 40mg — An intra-articular cocktail injection ( Ketoralac 15mg, Ropivacaine 1% 15ml, 0.9% Normal Saline 35ml, Adrenaline 1:1000 0.5ml, Stacort-A Triamcinolone Acetonide 40mg) will be injected into the surgical site after fracture fixation surgery.
  Arms: Intra-Articular Cocktail Injection
Drug: Ropivacaine HCL 1% 15ml — An intra-articular cocktail injection ( Ketoralac 15mg, Ropivacaine 1% 15ml, 0.9% Normal Saline 35ml, Adrenaline 1:1000 0.5ml, Stacort-A Triamcinolone Acetonide 40mg) will be injected into the surgical site after fracture fixation surgery.
  Arms: Intra-Articular Cocktail Injection
Drug: 0.9 % Normal Saline 35ml — An intra-articular cocktail injection ( Ketoralac 15mg, Ropivacaine 1% 15ml, 0.9% Normal Saline 35ml, Adrenaline 1:1000 0.5ml, Stacort-A Triamcinolone Acetonide 40mg) will be injected into the surgical site after fracture fixation surgery.
  Arms: Intra-Articular Cocktail Injection
Drug: Adrenaline 1:1000 0.5ml — An intra-articular cocktail injection ( Ketoralac 15mg, Ropivacaine 1% 15ml, 0.9% Normal Saline 35ml, Adrenaline 1:1000 0.5ml, Stacort-A Triamcinolone Acetonide 40mg) will be injected into the surgical site after fracture fixation surgery.
  Arms: Intra-Articular Cocktail Injection

SUMMARY:
The objective of this study is to demonstrate the safety and efficacy of an intra-articular analgesics cocktail injection for post-operative patella fracture fixation patients, by comparing post-operative pain relief and functional recovery among study subjects who received the injection and those who did not receive the injection. Secondary objective is to demonstrate the health economic effects of intra-articular analgesics cocktail injection by reducing length of hospital stay and reducing bed-stay related complications.

DETAILED DESCRIPTION:
This is a single-centre, double-blinded, randomised control trial that evaluates the efficacy of intra-articular analgesics cocktail injection in post-operative pain relief and functional recovery for fractured patella fixation patients. The recruited study subjects will be randomised to the two study groups respectively in a 1:1 randomisation ratio.

Patella is the largest sesamoid bone in the human body, it acts as the fulcrum of our knee extensor apparatus and is important during the gait cycle. Patella fracture commonly occurs after a fall on a flexed knee. Treatment can be conservative or surgical with open reduction and internal fixation. Patients often experience significant pain around the knee post-operatively, limiting their walking ability and hindering their rehabilitation. As a result, total hospital stay will be prolonged, leading to hospital stay-related morbidity and additional healthcare economic burden.

Previous studies have shown that the use of an analgesic cocktail injection in arthroplasty cases can significantly reduce early postoperative pain and provide better early motion. The cocktail regime is as follows for a unilateral joint:

Ketoralac 15mg Ropivacaine 1% 15ml 0.9% Normal Saline 35ml Adrenaline 1:1000 0.5ml Stacort-A Triamcinolone Acetonide 40mg Total Cocktail Volume ~50ml

After fracture fixation, patients in the intervention group will receive an intra-articular injection of the above analgesic cocktail, while patients in the control group will not receive an injection.

Herein this study, the investigators hope to demonstrate the safety and efficacy of an intra-articular analgesics cocktail injection for post-operative patella fracture fixation patients.

ELIGIBILITY:
Inclusion Criteria:

* acute patella fracture requiring open reduction and internal fixation;
* able to consent to surgery;
* pre-morbid able to ambulate

Exclusion Criteria:

* open fracture;
* polytrauma;
* previous knee arthroplasty;
* history of chronic pain,
* insulin-dependent diabetes mellitus, or peptic ulcer disease;
* chronic users of glucocorticoids, immunosuppressants, or immune-modulating agents, or of strong opioids (e.g.: morphine, fentanyl, hydromorphone, methadone, oxycodone, or meperidine);
* hepatitis B or C carrier;
* renal impairment (creatinine [Cr], >200 mmol/L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Pain as measured by Numerical Patient Reported Scale (NRPS) | Pre-op, Post-op Day 1 to 3
  Numerical Patient Reported Scale (NRPS), 0 (no pain) to 10 (worst pain imaginable)
Maximum Active Knee Flexion | At post-op Day 1 to 3
  The patient's Knee flexion is measured by a physiotherapist
Oral analgesics consumed | Post-operative 2 weeks period
  The level of the analgesic consumed (non-opioids, weak opioids, strong opioids), and the frequency of consumption
Tegner Lysholm Knee Score | Post-op Day 14
  The Lysholm Knee Score calculates and grades an overall score from 0 to 100 based on 8 domains: squatting, locking, pain, stair climbing, support, instability, and edema. Scores between 95 and 100 are regarded as exceptional, 84 and 94 as acceptable, 65 to 83 as fair, and less than 65 as poor.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Post-op Day 14
  The KOOS's five patient-relevant dimensions are scored separately: Pain (nine items); Symptoms (seven items); ADL Function (17 items); Sport and Recreation Function (five items); Quality of Life (four items). A Likert scale is used, and all items have five possible answer options scored from 0 (No problems) to 4 (Extreme problems), and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopaedic scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.
9-item Quality of Recovery Score (QoR-9 Score) | Post-op Day 1 to 3
  The QoR-9 has 9 questions evaluating the quality of recovery after surgery and anaesthesia. It is a patient-rated score ranging from 0 (worst) to 2 (best).

SECONDARY OUTCOMES:
Length of hospital stay | Through study completion, an average of 1 year
  The number of days the patient was hospitalised
Time to radiological bony union | Through study completion, an average of 1 year
  X-rays will be taken at different follow-up intervals (post-op 2 weeks, 6 weeks, 3 months, 6 months, 12 months). The X-rays will be assessed for bony union at the surgical site.
Incidence of Complications | Through study completion, an average of 1 year
  Complications such as fracture site infection, loss of reduction, non-union, and malunion will be assessed and recorded

CONTACTS AND LOCATIONS:
Overall Officials: Christian Fang, Principal Investigator — Dept of Orthopaedics and Traumatology, Queen Mary Hospital
Locations (1):
- Queen Mary Hospital, The University of Hong Kong, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Anonymized dataset to be included as supplementary data in the final publication
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: Additional information available upon reasonable request of principal investigator

REFERENCES:
- [Background] Baid M, Narula S, Manara JR, Blakeney W. Evolution in the Management of Patella Fractures. J Clin Med. 2024 Feb 29;13(5):1426. doi: 10.3390/jcm13051426. PMID 38592262
- [Background] Petrie J, Sassoon A, Langford J. Complications of patellar fracture repair: treatment and results. J Knee Surg. 2013 Oct;26(5):309-12. doi: 10.1055/s-0033-1353990. Epub 2013 Aug 16. PMID 23955187